CLINICAL TRIAL: NCT04873154
Title: Significance of CD133 Expression in Invasive Ductal Carcinoma of the Breast
Brief Title: CD133 Expression in Mammary Invasive Ductal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nagwa Abd El-Sadek Ahmed, Lecturer at Pathology Department, Faculty of Medicine, Sohag University, Sohag University
Other Study IDs: CD133, Breast Cancer
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
Keywords: CD133; IDC; Breast cancer progression
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background and Aim: Breast carcinoma is the most common type of cancer and the most common cause of cancer-related mortality among women worldwide. Cancer stem cells (CSCs) are thought to be responsible for tumor initiation, progression, dissemination and resistance to chemotherapy and radiotherapy. CD133 is a trans-membrane glycoprotein which is considered as a putative CSCs marker. It has been extensively used as a stem cell marker for normal and cancerous tissues. Emerging evidence suggests that CD133 may be a critical factor in tumor development, progression and metastasis. The aim of this study was to evaluate expression status of CD133 in invasive ductal carcinoma (IDC) of the breast and its role during breast cancer progression and to correlate its expression with some known clinicopathological parameters.

DETAILED DESCRIPTION:
Introduction:

Breast carcinoma is the most frequent malignant tumor in women worldwide comprising 30% on average of all cancers and the most likely cause of cancer-related deaths in women worldwide. In Egypt, according to the official statistics of the National Cancer Institute, Cairo University, breast carcinoma is the most prevalent cancer among women representing 35.1% of total cancer cases.

Breast carcinoma is currently regarded as a heterogeneous group of tumors with diverse morphology, behavior, outcome and response to therapy. In spite of advances in diagnosis and treatment of breast carcinoma, the clinical outcome remains unsatisfactory due to recurrence, metastasis or chemotherapy-resistance.

Cancer stem cells (CSCs) are recognized as a subpopulation of cancer cells that show the characteristics of normal stem cells. They are believed to possess the capacity to self-renewal and are responsible for tumor formation and progression. CSCs also promote tumor cell heterogeneity and metastasis. In addition, CSCs are thought to be more resistant to chemotherapy and radiotherapy. Given the significance of CSCs in tumor development, the identification and characterization of CSCs could lead to the development of directed therapies against these aggressive cells, hence more effective treatments for cancer.

Over recent years, CSCs have been described in different types of cancers including breast cancer. In the mammary gland, the microenvironment provides clues to control the behavior of epithelial stem and progenitor cells. Breast cancer stem cells (BCSCs) subpopulation was shown to express higher level of pro-invasive genes and had highly invasive properties.

With evidence forthcoming regarding the effects of the stroma and the microenvironment in breast tumor progression, several genes have also been reported to be associated with BCSCs. The phenomenon of epithelial-mesenchymal transition (EMT) is important discovery during progression of breast carcinoma and explanation for their ability to invade and to colonize other parts of the body. With all these knowledge, targeting BCSCs for breast carcinoma treatment was demanded.

CD133, also known as prominin-1, is a member of pentaspan trans-membrane glycoproteins, frequently expressed on multipotent progenitor cells, including immature hematopoietic stem and progenitor cells. CD133 is a putative CSCs marker; it has been extensively used as a stem cell marker for normal and cancerous tissues. CD133 expressing cells possessing stem cell-like characteristics including self-renewal, high proliferation and drug resistance substantiating a tumorigenic role of CD133-expressing cells. It also plays a role in cell differentiation, proliferation and apoptosis.

Emerging evidences suggest that CD133 may be a critical factor in tumor development, progression and metastasis. CD133-positive CSC showed increased expression levels of CXCR4 which is a critical protein for the adhesion and/or migration of tumor cells, indicating an important role of CD133 in tumor cells migration and tumor invasion. CD133 is used as a diagnostic and prognostic marker which is overexpressed in various neoplasms. In breast cancer, its overexpression confers a poor prognosis. Increasing clinical evidence has confirmed that it is involved in breast cancer progression. CD133 is a promising marker for the identification of CSC in breast cancer subtypes including aggressive HER2+ and triple-negative classes.

Aim of This Work:

The aim of this study is to

1. Detect the immunohistochemical expression of CD133 in mammary invasive ductal carcinoma (IDC) and to correlate its expression with some known clinicopathological parameters.
2. Correlate the IHC expression of CD133 with some known clinicopathological parameters in mammary IDC.

ELIGIBILITY:
Inclusion Criteria:• Inclusion criteria: Patients with IDC and underwent mastectomy or excisional biopsy of breast mass.

-

Exclusion Criteria

* Patients received pre-operative chemotherapy or radiotherapy.
* Patients with insufficient clinical data.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: • Patients: Fifty specimens of IDC obtained from patients who underwent mastectomy in General Surgery Department of Sohag Faculty of Medicine according to local Ethical Committee regulations, to be examined in the Pathology Laboratory of the same faculty.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
1. Detect the immunohistochemical expression of CD133 in mammary invasive ductal carcinoma (IDC) and to correlate its expression with some known clinicopathological parameters. | 1 month

SECONDARY OUTCOMES:
2. Correlate the IHC expression of CD133 with some known clinicopathological parameters in mammary IDC. | 1 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt